CLINICAL TRIAL: NCT04514094
Title: Effectiveness of Silver Diamine Fluoride in Arresting Early Childhood Caries: Randomized Controlled Clinical Trial
Brief Title: Silver Diamine Fluoride Effectiveness Versus Atraumatic Restorative Treatment in Arresting ECC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDF Trials
Record Dates: First submitted 2020-08-13; First posted 2020-08-14 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Early Childhood Caries
MeSH Terms: interventions — silver diamine fluoride

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silver Diamine Fluoride (Experimental): * Gross debris will be removed with cotton pellets to allow better SDF contact with denatured dentin.
  * Cotton rolls will be used to protect surrounding gingival tissues and mucous membranes to avoid pigmentation or irritation.
  * Affected tooth surfaces will be dried with a gentle flow of air.
  * 1-2 drops only of SDF will be used for the whole visit.
  * SDF will then be directly applied to affected tooth surfaces only using a micro sponge brush.
  * At least one minute will be needed to allow drying of SDF.
  * Excess SDF will finally be removed with cotton rolls to minimize systemic absorption.
  * When possible, isolation will be continued for up to three minutes.
  * After 2-4 weeks: reapplication will be done only to lesions that do not appear arrested (dark and hard).
  Interventions: Drug: SDF
- Atraumatic Restorative Treatment (Active Comparator): Caries removal by hand instruments with care not to expose the pulp.
  * Maximum excavation from the periphery of lesions will be done, to minimize leakage at the restoration margins.
  * Cotton roll isolation will then be carried out.
  * Cavities will be restored by glass ionomer cement.
  * Hand pressure should be applied by a gloved and petroleum jelly coated finger, then, excess material will be removed.
  Interventions: Procedure: ART

INTERVENTIONS:
Drug: SDF — SDF promotes enamel and dentin remineralization, as well as inhibit the growth of cariogenic bacteria. the Food and Drug Administration (FDA) approved SDF as a device for reducing tooth sensitivity in the USA.
  Other Names: Silver Diamine Fluoride
  Arms: Silver Diamine Fluoride
Procedure: ART — The ART technique involves caries excavation by hand instruments only with care to avoid pulp exposure. Such excavation is mainly from the periphery of the lesion to achieve a good seal of the restoration and minimize leakage. The tooth is then restored by glass ionomer cement.
  Arms: Atraumatic Restorative Treatment

SUMMARY:
The study was conducted to evaluate the effectiveness of the biannual application of 38% silver diamine fluoride in arresting early childhood caries when compared to atraumatic restorative treatment.

DETAILED DESCRIPTION:
Owing to the virulent nature of early childhood caries (ECC) and its consequences if left untreated, immediate intervention is indicated to control the condition.

Barriers to intervention as young age, uncooperative patient behavior and lack of access to dental care are however, very common. The use of silver diamine fluoride as an anticaries agent is of growing popularity worldwide due to its promising results, safety of use, ease of application and relatively low cost. Further research is still required in order to provide evidence-based recommendations regarding the use of SDF in arresting early childhood caries. Purpose: To evaluate the effectiveness of biannual application of 38% silver diamine fluoride in arresting early childhood caries when compared to atraumatic restorative treatment.

ELIGIBILITY:
Inclusion Criteria:

* For children:

  1. Healthy children.
  2. Age range 2-5 years.
  3. Informed consent (Appendix I)

For teeth:

* Teeth with active dentin lesions corresponding to ICDAS II score 5 and 6.
* Teeth having lesions that are considered active according to ICDAS II activity criteria for coronal primary caries.

Exclusion Criteria:

* For children:

  1. Children with systemic diseases.
  2. Children with reported allergy to silver or to any other component in the materials used.
  3. Children unable to return for recall visits.

For teeth:

* Clinical or radiographic signs of pulpal involvement.(pain, abscess, sinus, obvious discoloration, premature hypermobility, internal or external root resorption).
* Teeth with inactive lesions.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2019-08-23 (Actual)

PRIMARY OUTCOMES:
change in clinical success/failure rate | at 6 and 12 months
  Treated teeth in both groups will be evaluated for clinical success in each follow up appointment. The number of clinically successful/failed teeth will be recorded in

SECONDARY OUTCOMES:
Duration of the intervention visit | During the procedure
  time spent during each intervention appointment was calculated in seconds
Patient Satisfaction | after the 4th week
  using a 4-item, 5-level, Likert-scale questionnaire o assess feelings about the application procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt